CLINICAL TRIAL: NCT03186001
Title: The Impact of Botulinum Toxin Injection in the Frontalis on Brow Height and Morphology: A Randomized Trial
Brief Title: Frontalis Botulinum Toxin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, samer jabbour, M.D., St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USJ-06
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Browlift
Keywords: frontalis; frontal line; glabellar line; botulinum toxin; abobotulinum
MeSH Terms: interventions — abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- v shape (Experimental): Technique 1Lateral orbicularis and corrugator injections: 5 equally spaced injections will be placed intramuscularly into the orbicularis under the lateral eyebrow starting lateral to the level of the lateral limbus and extending to the level of the inferior orbital rim. In addition, 2 injections will be placed 1cm apart into the corrugator starting at the medial brow and extending laterally. Then 5 equally spaced injections, in a V pattern will be placed in the frontalis. The first injection between the medial brows, 2 injection 1cm below the hairline at the level of the lateral canthus and one injection equidistant to medial and lateral injection.
  Interventions: Drug: Abobotulinum toxin A
- middle frontalis (Experimental): : Lateral orbicularis and corrugator injections: 5 equally spaced injections will be placed intramuscularly into the orbicularis under the lateral eyebrow starting lateral to the level of the lateral limbus and extending to the level of the inferior orbital rim. In addition, 2 injections will be placed 1cm apart into the corrugator starting at the medial brow and extending laterally. Then 5 equally spaced injections, in a straight pattern will be placed in the frontalis. One injection in the middle of the forehead, one on the same level of the lateral canthus and one between them.
  Interventions: Drug: Abobotulinum toxin A
- high frontalis (Experimental): : Lateral orbicularis and corrugator injections: 5 equally spaced injections will be placed intramuscularly into the orbicularis under the lateral eyebrow starting lateral to the level of the lateral limbus and extending to the level of the inferior orbital rim. In addition, 2 injections will be placed 1cm apart into the corrugator starting at the medial brow and extending laterally.Then 5 equally spaced injections, in a straight pattern 1 cm below the hairline will be placed in the frontalis. One injection in the middle of the forehead, one on the same level of the lateral canthus and one between them.
  Interventions: Drug: Abobotulinum toxin A

INTERVENTIONS:
Drug: Abobotulinum toxin A — The purpose of this study is to describe two safe and reproducible techniques upper face botulinum toxin injection. It will also describe the effect of both techniques on the eyebrow shape and height using quantitative, objective measurements and subjective scales

SUMMARY:
The botulinum toxin was first identified in the late 19th century(1). With its 40 different subtype this toxin is produced mainly by the gram positive anaerobic bacteria Clostridium Botulinum(2). This neurotoxin has great affinity to the neuro muscular junction preventing neurotransmitter release in the synaptic space of acetylcholine(3). The first clinical use was reported by Alan Scott in 1980(4). The most commonly used subtype is toxin A commercially found as BOTOX (onabotulinumtoxinA, Allergan, approved by FDA in 1989), Dysport (abobotulinumtoxinA, Medicis, approved by FDA in 2009) and Xeomin (incobotulinumtoxinA, Merz, approved by FDA in 2010). As for other commercial toxins botulinum neurotoxin serotype B product (MYOBLOC™). Neurotoxin Blast generally 12-15 weeks compared to 3-6 month for neurotoxin A. the FDA approved its use for strabismus in 1989(5), blepharospasm and hemifacial spasm in 1990(6,7), cervical dystonia in 2000(8), glabella in 2000, hyperhidrosis in 2004(9), chronic migrane and detrusor overactiviy in 2014. Other off-label uses have emerged like lanyngeal dysponia, chronic pain etc… (10). Multiple studies with a reduced number of patients have aimed to quantify the effect of botulinum toxin on brow higth. Some studies used injections only to the lateral part of the orbicularis,while others added a corrugator injection. We aimed in this study to compare a known techniques in brow lifting and associanting that with 2 frontalis injection techniques. The main objective is to evaluate the shape of the brow and the elevation in multiple brow landmarks before and after the injection and to see if the frontalis botulinum bloc causes brow ptosis

DETAILED DESCRIPTION:
Botulinum toxin:

This toxin has been used clinically since 1989 with label (8) and off-label techniques(3).

This is a becoming a routine procedure for men and women with little side effects.

Brow lifting The ideal brow position is always an issue in plastic surgery(12). When face ages, the brow descends. Many approaches to a brow elevation are described in the literature. The first surgical approach is through a coronal incision(13), then came the temporal incision(14) and the direct approach(15), and finally the endoscopic approach(16). Non-surgical methods include radiofrequency(17), percutaneous sutures and botulinum toxin(11).

Standardized measure Anteroposterior pictures will be taken at rest pre and post injection. Using photoshop 7 brow landmarks will be measured to the midpupillary line.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive 30 female patients presenting to our clinic for brow lifting with botulinum toxin will be randomized to receive one of the two injection techniques
2. 30 Years to 60 Years
3. Female

Exclusion Criteria:

1. Patients with previous periorbital/forehead surgery
2. Patients who plucked the upper eyebrow margin
3. Patients with eyebrow tatoos
4. Patients with upper face botulinum toxin injection in the past 12 months
5. Patients with resorbable upper face fillers injection in the past 12 months
6. Patients with previous permanent upper face fillers injection
7. Pregnant patients
8. Lactating patients
9. Patients with preexisting neuromuscular conditions (myasthenia gravis, Eaton Lambert syndrome)
10. Patients using medication that could potentiate the effect of botulinum (ex: aminoglycoside antibiotics)
11. Patients with sensitivity to botulinum toxin or human albumin

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective assessment | 2 weeks
  Objective assessment will be done on anteroposterior views of pre-and-post injection photographs. The mid pupillary line will be drawn and the eyebrow vertical height will be measured from this line to the upper border of the brow at seven horizontal points: the most medial aspect of the eyebrow, medial canthus, and medial limbus, mid pupil, lateral limbus, lateral canthus, and most lateral eyebrow.

SECONDARY OUTCOMES:
1-Investigators Global Aesthetic Improvement Scale | 2 weeks
  Improvement in Overall appearance of the upper face, as assessed by the 3 investigators (2 plastic surgeons and 1 dermatologist) using the Global Aesthetic Improvement Scale (GAIS). GAIS will be completed based on photographic assessment comparing post-treatment photos taken at day 15 post intervention to baseline photos (the lower eyelids and lower face will be cropped), to assess overall aesthetic improvement. The GAIS is a 5-point scale (1-5) as follows:
  1. Very Much Improved: optimal cosmetic results
  2. Much Improved: marked improvement in appearance from initial condition but not completely optimal
  3. Improved: obvious improvement in appearance from initial condition but additional treatments are advised
  4. No Change: the appearance is the same as the original condition
  5. Wose: the appearance is worse from the original condition
2-Patient satisfaction | 2 weeks
  Patient satisfaction will be determined by a questionnaire completed at 15 days post-treatment. Subjects will indicate how satisfied they are on a 4-point scale (1-4) as follow:
  1. Very Satisfied
  2. Satisfied
  3. Dissatisfied
  4. Very Dissatisfied.
3-Brow Positioning Scale | 2 weeks
  subjective evaluation using a photonumeric validated scale for eye brow positioning (evaluated by 2 plastic surgeons and 1 dermatologist) using pre and post injection photographs (taken at day 15 and 30) as follow: 0-Youthful, refreshed look and high-arch eyebrow
  1. Medium-arch eyebrow
  2. Slight arch of the eyebrow
  3. Flat arch of the eyebrow, visibility of folds, and tired appearance
  4. Flat eyebrow with barely any arch, marked visibility of folds, and very tired appearance
4-Forehead Lines Scale: | 2 weeks
  subjective evaluation using a photonumeric validated scale for forehead lines at rest (evaluated by 2 plastic surgeons and 1 dermatologist) using pre and post injection photographs (taken at day 15 and 30) as follow: 0-None
  1. Minimal
  2. Moderate
  3. Deep
  4. Extreme
5-Glabellar Lines Scale | 2 weeks
  subjective evaluation using a photonumeric validated scale for glabella lines at rest (evaluated by 2 plastic surgeons and 1 dermatologist) using pre and post injection photographs (taken at day 15) as follow: 0-No glabella lines
  1. Mild glabella lines
  2. Moderate glabella lines
  3. Severe glabella lines
  4. Very severe glabella lines

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Joseph University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jabbour SF, Awaida CJ, ElKhoury JS, Rayess YA, Makhoul RB, Kechichian EG, Nasr MW. The Impact of Upper Face Botulinum Toxin Injections on Eyebrow Height and Forehead Lines: A Randomized Controlled Trial and an Algorithmic Approach to Forehead Injection. Plast Reconstr Surg. 2018 Nov;142(5):1212-1217. doi: 10.1097/PRS.0000000000004836. PMID 30102667